CLINICAL TRIAL: NCT03281850
Title: The GLOWING Study: Growing Life, Optimizing Wellness 2
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 206846
Record Dates: First submitted 2017-09-07; First posted 2017-09-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Urine collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study will help us learn more about how maternal health can influence child health.

DETAILED DESCRIPTION:
This study follows people who are healthy and less than 36 weeks pregnant to see how the mother's health can impact their child's growth and development. Up to 300 people including the mother and their future child will be a part of this study. The study will follow the child until they are two years of age.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pregnancy BMI 18.5-45
* Singleton pregnancy
* at least 18 years of age
* conceived without assisted fertility treatments

Exclusion Criteria:

* Preexisting medical conditions (e.g. DM, GDM, CRF, HTN, pre-eclampsia or eclampsia, malignancies, seizure disorder, lupus, serious psychiatric disorders)
* sexually transmitted diseases
* medications during pregnancy known to influence fetal growth
* smoking, alcohol drinking or drug use during pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective longitudinal cohort of 150 dyads (pregnant women and offspring)
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Determine energy expenditure in children | 2 years
  Using stable isotope techniques to determine energy expenditure
Determine fat oxidation in children | 2 years
  Using stable isotope techniques to determine fat oxidation

CONTACTS AND LOCATIONS:
Overall Officials: Aline Andres, PhD, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Diaz EC, Williams DK, Cotter M, Sims CR, Wolfe RR, Andres A, Borsheim E. Breastfeeding duration modifies the association between maternal weight status and offspring dietary palmitate oxidation. Am J Clin Nutr. 2022 Aug 4;116(2):404-414. doi: 10.1093/ajcn/nqac097. PMID 35404455